CLINICAL TRIAL: NCT06658314
Title: Comparison of Kinesiotaping and Graded Exposure Therapy on Kinesiophobia in Post-Mastectomy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RiphahIU Madiha Bashir
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Post-mastectomy Pain Syndrome
Keywords: Kinesiophobia; Kinesiotaping; Graded exposure therapy; Post-mastectomy patients
MeSH Terms: conditions — Kinesiophobia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: interventional group 1(Kinesiotaping) (Active Comparator): Kinesiotape will be applied by using two I-bands application technique. It will be applied once a week for 3 to 5 days and total time period of 3 weeks.
  Interventions: Other: Experimental interventional group 1(Kinesiotaping)
- Experimental :interventional group II (Graded exposure therapy) (Experimental): Graded exposure therapy consists of set of exercises, performed for 3 weeks with 3 sessions per week. Each exercise protocol has 5 to 10 repetitions per day.
  Interventions: Other: Experimental interventional group II (Graded exposure therapy)

INTERVENTIONS:
Other: Experimental interventional group 1(Kinesiotaping) — Kinesiotape will be applied by using two I-bands application technique:
  Short band: to apply this ask the patient to move your arm behind her back as much as possible, then apply kinesiotape at the anterior glenohumeral joint.
  Longer band: to apply this ask the patient to horizontal adduct her arm as much as possible, than apply kinesiotape targeting the posterior side of glenohumeral joint.
  Apply both these band with paper-off stretch for 3-5 days or as depending upon skin sensitivity and tape adherence.
  Kinesiotape will be applied once a week for total time period of 3 weeks.
  Arms: Experimental: interventional group 1(Kinesiotaping)
Other: Experimental interventional group II (Graded exposure therapy) — First week: gentle arm raises with 10 repetitions/day, slow and controlled stretch 25 to 50% force with 5 repetitions, passive internal and external rotations (with towel) with 5 repetitions each/day.
  Second week: overhead arm raises (wall climbing) with 10 repetitions/day, pendulum exercises 10 repetitions/day, cross arm stretches 5 repetitions/day, active internal and external rotations with 5 repetitions each/day.
  Third week: resistance exercises (initially with minimum weight or manual resistance), scapular squeezes 10 repetitions/day, gentle chest stretches 5 repetitions/day and gentle stretch with 75 to 100 % force 5 repetitions each/day.
  Arms: Experimental :interventional group II (Graded exposure therapy)

SUMMARY:
The aim of this research is to compare the effect of Comparison of Kinesiotaping and Graded exposure therapy on Kinesiophobia in Post-Mastectomy patients. The sample size was 30. The subjects were divided in two groups, 15 subjects in kinesiotaping group and 15 in graded exposure therapy group. Study duration was of 1 year. Sampling technique applied was nonprobability Convenience sampling technique. Patients had recently undergone mastectomy procedure age between 30 to 60 years and mean Tempa- 11 score of >23 were included. Tools used in the study are Tempa -11 for kinesiophobia, NPRS for Pain, SPADI for Functional outcome measure. Data was be analyzed through SPSS 26.

DETAILED DESCRIPTION:
Mastectomy is a procedure performed as a part of treatment for breast cancer, which entails removal of entire breast tissue. Breast cancer is a condition where abnormal cells in the breasts proliferate and eventually develop tumor. It is the most prevalent form of cancer accounting for 23% of all the newly diagnosed cancers. There are several types of mastectomy procedures including complete mastectomy, radical mastectomy and modified radical mastectomy. After mastectomy, many possible complications and side effects can occur including seroma, lymphedema, pain, restricted range of motion, kinesiophobia, infection etc. and all these complications required special care and treatment to improve patient's quality of life. Breast cancer survivor often develop fear of movement called kinesiophobia either due to pain or other psychological factors. It is the excessive, irrational, and debilitating fear of movement or physical activity. This fear of movement is linked to a feeling of susceptibility to injury from movement. As a result of using the painful area less due to the fear of increased pain from movement, acute pain can develop into persistent and chronic pain that in return increase hospital stay and decrease quality of life which increase the financial burden on individual. According to the recent studies kinesiophobia is one of the parameters found in post-mastectomy patients with mean Tempa -11 score of 24 in Pakistani populations.

Post mastectomy complications are mostly manageable, and studies show significant improvement in patient's symptoms. Shoulder disability, pain and ROM are addressed in many studies but managing kinesiophobia in early stages after mastectomy still needs to be further discussed

ELIGIBILITY:
Inclusion Criteria:

* Females
* Age between 30-60 years.
* Post-Mastectomy patients (not more than 4 weeks).
* Tempa -11 score >23.

Exclusion Criteria:

* Any shoulder dislocations/fracture.
* Any known neurological impairments i.e. radiculopathy
* Bilateral mastectomy
* Known Cardiac issues
* Patients undergoing chemotherapy
* Any known allergies to kinesiotaping

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 32 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-06-19 (Actual)

PRIMARY OUTCOMES:
Tempa-11 Scale | Kinesiophobia will be assessed at baseline to 3rd week
  Tempa-11 Scale is used to measure Kinesiophobia. This questionnaire has 11 items with the total score of 44, 11 being the lowest possible score and 44 being the highest

SECONDARY OUTCOMES:
Numeric Pain Rating Scale | Pain will be assessed at baseline to 3rd week
  Numeric pain rating scale is used to assess pain. Numeric pain rating scale is a 11-item scale comprising usually of horizonal or vertical line with 0 to 10 ratings between the two extremes.
SPADI | it will be assessed at baseline to 3rd week
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire that consists of two main items, one for pain and the other for functional activities. The pain dimension consists of five questions regarding the severity of an individual's pain. Functional activities are assessed with eight questions designed to measure the degree of difficulty an individual face during various activities of daily living that require upper-extremity use.

CONTACTS AND LOCATIONS:
Overall Officials: Aisha Razzaq, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Fauji Foundation Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No